CLINICAL TRIAL: NCT06345300
Title: Liposomal Irinotecan，Oxaliplatin, 5-Fluorouracil/Calcium Folinate in Combination With Camrelizumab for Borderline Resectable Pancreatic Cancer: a Prospective, Exploratory Study
Brief Title: NALIRIFOX in Combination With Camrelizumab for BRPC: a Prospective, Exploratory Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4309
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-12

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: Liposomal Irinotecan; borderline resectable pancreatic cancer
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab (Experimental): Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab
  Interventions: Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab
- Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate (Experimental): Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate
  Interventions: Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate

INTERVENTIONS:
Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab — The treatment regimen for this study is as follows:
  Intravenous infusion of Oxaliplatin at a dose of 85mg/m2 for 2 hours or according to clinical practice at the research center;
  Intravenous infusion of liposomal Irinotecan at a dose of 60mg/m2 for 90 minutes (±30 min);
  Intravenous drip of Calcium folinate at a dose of 400mg/m2 for 30 minutes or according to clinical practice at the research center;
  Intravenous infusion of 5-Fluorouracil at a dose of 2400mg/m2 (infused for 46-48 hours or according to clinical practice at the research center);
  Camrelizumab at a fixed dose of 200mg, administered via intravenous drip, with each infusion lasting no less than 30 min and no more than 60 min. Administered on day 1 of every 2-week cycle (d1, q2w).
  Each treatment cycle is 14 days, and all drugs are administered on day 1.
  Other Names: NALIRIFOX+PD-1
  Arms: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab
Drug: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate — The treatment regimen for this study is as follows:
  Intravenous infusion of Oxaliplatin at a dose of 85mg/m2 for 2 hours or according to clinical practice at the research center;
  Intravenous infusion of liposomal Irinotecan at a dose of 60mg/m2 for 90 minutes (±30 min);
  Intravenous drip of Calcium folinate at a dose of 400mg/m2 for 30 minutes or according to clinical practice at the research center;
  Intravenous infusion of 5-Fluorouracil at a dose of 2400mg/m2 (infused for 46-48 hours or according to clinical practice at the research center); Each treatment cycle is 14 days, and all drugs are administered on day 1.
  Other Names: NALIRIFOX
  Arms: Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate

SUMMARY:
The aim of this study is to assess the efficacy and safety of Liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate in combination with Camrelizumab for patients with borderline resectable pancreatic cancer

DETAILED DESCRIPTION:
This study plans to include 40 patients with borderline resectable pancreatic cancer who are evaluated by a multidisciplinary team (MDT). These patients will receive 3 cycles of neoadjuvant therapy before surgery. The immunotherapy combination chemotherapy regimen consists of liposomal Irinotecan, Oxaliplatin, 5-Fluorouracil/Calcium folinate, and Camrelizumab, with a 14-day dosing cycle. The chemotherapy regimen consists of liposomal Irinotecan, Oxaliplatin, and 5-Fluorouracil/Calcium folinate.

Clinical tumor imaging evaluation will be conducted based on the RECIST 1.1 criteria after the completion of neoadjuvant therapy. The MDT will assess whether patients are eligible for surgery based on the imaging results. The criteria for operability include: no evidence of implantation metastasis during laparoscopic exploration, absence of new metastatic lesions, and the tumor's relationship with blood vessels meeting the criteria for R0/R1 resection.

Patients eligible for surgery will undergo pancreatic cancer surgery 4-6 weeks later. Postoperative treatment will be determined by the researchers based on the neoadjuvant treatment effectiveness and the patients'actual conditions. Imaging evaluations will follow the standard diagnostic and treatment guidelines for pancreatic cancer.

For patients deemed ineligible for surgery, the subsequent treatment plan will be determined by the researchers based on the neoadjuvant treatment effectiveness and the patients' actual conditions

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, both males and females are eligible.
2. Histologically or cytologically confirmed pancreatic cancer (originating from pancreatic duct epithelium) assessed by Multidisciplinary Team (MDT) as potentially resectable pancreatic cancer. (According to CSCO guidelines 2022, potentially resectable pancreatic cancer is defined as:Tumor involvement with the portal vein-mesenteric vein >180° or contact ≤180° with irregular vein contour or vein thrombosis, but can be completely resected and safely reconstructed; tumor involvement with the inferior vena cava;(Tumor involving the pancreatic head/uncinate process) Tumor involvement with the hepatic artery distal to the celiac trunk, with no involvement of the celiac trunk or the origin of the left or right hepatic artery, can be completely resected and safely reconstructed; tumor involvement with the mesenteric artery ≤180°; tumor involvement with variant arteries (such as accessory right hepatic artery, replaced right hepatic artery, replaced common hepatic artery, etc.).(Tumor involving the body and tail of the pancreas) Tumor involvement with the mesenteric artery ≤180°; tumor involvement with the celiac trunk ≤180°).
3. No prior treatment with local or systemic anti-tumor therapy, including chemotherapy, radiation therapy, targeted therapy, or immunotherapy.
4. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Expected survival of ≥12 weeks.
7. Adequate organ function as follows (no use of any blood components, growth factors, leukocyte-boosting agents, platelet-boosting agents, or anemia correction drugs within 14 days prior to the first use of study medication):

   1. Absolute neutrophil count (ANC) ≥1.5×10*9/L;
   2. Platelets ≥85×10*9/L;
   3. Hemoglobin ≥90 g/L;
   4. Serum albumin ≥30 g/L;
   5. Total bilirubin ≤2.0 × upper limit of normal (ULN) (patients with biliary obstruction after biliary drainage ≤2.5 × ULN), AST and ALT ≤3.0 × ULN (patients with liver metastasis ≤5 × ULN);
   6. Creatinine clearance > 60 mL/min;
   7. Activated partial thromboplastin time (APTT) and International Normalized Ratio (INR) ≤1.5 × ULN (patients taking stable doses of anticoagulants such as low molecular weight heparin or warfarin and INR within the expected therapeutic range of the anticoagulant can be included).
8. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days before enrollment and agree to use appropriate contraception during the observation period and up to 8 weeks after the last administration of the study drug; for males, they must have undergone surgical sterilization or agree to use appropriate contraception during the observation period and up to 12 weeks after the last administration of the study drug.
9. Participate in the study and signing of an informed consent form.

Exclusion Criteria:

* Participants who meet any of the following criteria will not be allowed to enter this study:

  1. Pancreatic cancer originating from non-pancreatic ductal epithelium, including pancreatic neuroendocrine tumors, pancreatic acinar cell carcinoma, pancreatic embryonal carcinoma, solid pseudo-papillary tumors.
  2. Patients with central nervous system metastasis.
  3. Severe gastrointestinal dysfunction (with bleeding, inflammation, obstruction, or diarrhea classified as grade 1 or higher).
  4. Existence of grade 3 or 4 peripheral neuropathy.
  5. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring drainage.
  6. Uncontrolled systemic infection (viral, bacterial, and fungal).
  7. Allergy to previous use of erlotinib liposomes, other liposomal products, oxaliplatin, 5-fluorouracil, calcium folinate, or any component of the mentioned products.
  8. Allergy to monoclonal antibodies, camrelizumab, or any component of the investigational drug.
  9. Use of any investigational drug within 4 weeks prior to the first use of the investigational drug in this study.
  10. Receipt of the last dose of anticancer therapy (including radiotherapy) within 4 weeks prior to the first use of the investigational drug.
  11. Underwent major surgery within 4 weeks prior to the first use of the investigational drug.
  12. Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study or follow-up of an interventional clinical study.
  13. Participants with poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or higher heart failure; (2) unstable angina pectoris; (3) myocardial infarction within the past year.
  14. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) or hepatitis C (positive anti-HCV or HCV-RNA above the detection limit of the assay).
  15. Diagnosed with any other malignant tumor within 5 years prior to the first use of the investigational drug, excluding malignant tumors with low risk of metastasis and death (5-year survival rate > 90%), such as adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix.
  16. Pregnant or lactating women.
  17. Participant judged by the investigator to have other factors that may necessitate premature termination of the study, such as the presence of other serious diseases (including mental illnesses) requiring concurrent treatment, or family or social factors that may affect participant safety or data collection in the study.
  18. Other factors deemed by the investigator to make the participant unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 years
  Defined as the proportion of subjects with R0 resection assessed postoperatively

SECONDARY OUTCOMES:
Event free survival (EFS) | 1.5 years
  The time from randomization to the occurrence of any of the following events, whichever comes first:
  Radiographic tumor progression evaluated according to RECIST 1.1 criteria. Tumor recurrence assessed by imaging, including local recurrence or distant metastasis.
  Death due to any cause.
Overall survival (OS) | 2 years
  The time from the initiation of the first dose of medication in a patient to death from any cause.
Objective Response Rate(ORR) | 2year
  The proportion of patients with a confirmed complete response or partial response using RECIST 1.1
Disease Control Rate（DCR） | 2 years
  The proportion of patients with a best overall response of confirmed complete or partial response, or stable disease (CR+ PR + SD)
Safety and tolerability by incidence, severity and outcome of adverse events | 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijin, China